CLINICAL TRIAL: NCT03145012
Title: Histamine Receptor 2 Antagonists as Enhancers of Anti-Tumour Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SAIL-002
Record Dates: First submitted 2017-04-26; First posted 2017-05-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Cancer; Immunity; Peripheral Blood Mononuclear Cells; Ranitidine
MeSH Terms: conditions — Neoplasms | interventions — Ranitidine

STUDY DESIGN:
Intervention Model Description: Healthy individuals will be asked to take ranitidine for 6 weeks to determine the effect on peripheral blood immune cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): This is a one arm study in which all individuals receive the treatment; therefore there is no allocation or randomization.
  Thirty subjects will receive ranitidine to a maximum of 900 mg/day in 2 daily doses for 6 weeks. The dosage target is 8 mg/kg/day, but the range of ranitidine intake will be between 7.5- 9 mg/kg/day. This is due to the formulation of the tablets, sold as 75, 150, and 300mg tablets. The ranitidine will be taken orally.
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Ranitidine — Thirty subjects will receive Ranitidine to a maximum of 900 mg/day in 2 daily oral doses for 6 weeks. The dosage target is 8 mg/kg/day, but the range of ranitidine intake will be between 7.5- 9 mg/kg/day. This is due to the formulation of the tablets, sold as 75, 150, and 300mg tablets.
  Other Names: Zantac

SUMMARY:
The immune response against tumors can be highly effective in preventing tumor development, growth and metastasis under certain circumstances. However, tumor associated immune suppression can profoundly limit the impact of natural tumor immunity and also reduce the effectiveness of tumor immunotherapy strategies.

A major component of tumor associated immune suppression is mediated by myeloid cells, especially the monocytic subset of myeloid derived suppressor cells (MDSC). In recent studies that were conducted through a CCSRI Innovation grant, the investigators discovered that oral treatment of mice with the commonly used histamine receptor 2 (H2) antagonists ranitidine or famotidine inhibits both primary breast tumor development and metastasis, in three distinct mouse tumor models and reduces the numbers of monocytic MDSC. These findings have enormous potential to aid in effective cancer immunotherapy and may have immediate implications for cancer patients.

The objective of this investigation is to determine whether treatment with the H2 receptor antagonist ranitidine alters immune suppression, through modulation of immune cell populations.

The investigators will examine peripheral blood monocyte, neutrophil and NK cell numbers, subsets and activation status from healthy volunteers treated for 6 weeks with daily oral ranitidine.

Ranitidine is widely available and used over the counter in Canada. These drugs are widely recognized as safe, well tolerated and have very few side effects. It has been suggested that among the general population, over 10% of those over the age of 65 take such medications on a regular basis for relief against gastrointestinal discomfort. The outcome of pre-clinical studies in mice warrant further investigation into transferability to humans.

If the outcome of the current proposal proves to be viable, then these drugs could provide a safe method to reduce tumor associated immunosuppression with broad implications, both for current cancer patients and for those at high risk of developing cancer. Further to this, the outcome of our proposal may provide a new strategy for improving the effectiveness of T-cell mediated immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years old, all sexes or genders
* Veins acceptable for blood draw
* Able to provide informed consent
* eGFR > 90 mL/min/1.73m2
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG, urinalysis). Clinical laboratory values within stated normal range; if not within this range, they must be without clinical significance
* Female volunteers who are of childbearing potential that agree to use of the accepted contraceptive regimens from at least 21 days prior to the first administration of study drug, during the study, and for at least 30 days after the last dose of study drug
* Female volunteers who are postmenopausal (no menses for at least 1 year, or surgically sterile

Exclusion Criteria:

* Use of ranitidine for greater than 1 week within 6 months of starting the study
* Medical requirement for ranitidine use
* Current or past diagnosis of: porphyria, cancer, immune deficiency disorder
* Active infection at the time of screening
* Known liver, hematologic, renal disease
* Past history of allergic reaction to ranitidine or past history of hypersensitivity to any ingredient in the formulation or past history of hypersensitivity to other drugs
* Pregnant, planning to be pregnant, or breastfeeding during the study period
* Weight (kg) exceeds 109kg

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Intra-individual frequency and function of immune cell subsets | Frequency and function were calculated as the values at 6 wks after treatment compared to the values at baseline.
  To determine the effect of histamine 2 receptor antagonists on immune cell function in healthy humans. Frequency and function of B cell, T cell, monocyte, NK cell and MDSC cells will be assessed by flow cytometry and ELISPOT.

SECONDARY OUTCOMES:
Inter-individual frequency and function of immune cell subsets | Frequency and function were calculated as the values at 6 wks after treatment compared to the values at baseline.
  To determine the effect of histamine 2 receptor antagonists on immune cell function cross-sectionally. B cell, T cell, monocyte, NK cell and MDSC cells will be assessed by flow cytometry and ELISPOT.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Barrett, MD/PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD with other researchers.